CLINICAL TRIAL: NCT07114367
Title: An Open-Label, Multicenter, Monotherapy, Dose-Escalation, Phase 1 Clinical Trial of NB02 (Posseltinib) in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: NB02(POSELTINIB) Monotherapy in R/R Non-Hodgkin's Lymphoma
Acronym: POTENTIAL-M
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NOBO Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB02-L02
Record Dates: First submitted 2025-07-03; First posted 2025-08-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Hodgkin Lymphoma (NHL)
Keywords: Relapsed; Refractory; Lymphoma; NHL; FL; MCL; MZL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma | interventions — poseltinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NB02 (Poseltinib) (Experimental): Dose Level 1 Dose Level 2 Dose Level 3
  Interventions: Drug: NB02 (Poseltinib)

INTERVENTIONS:
Drug: NB02 (Poseltinib) — Dose Level 1, Dose Level 2, Dose Level 3

SUMMARY:
This trial is an open-label, multicenter, monotherapy, dose-escalation, phase 1 clinical trial to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of NB02 (posseltinib) in patients with relapsed/refractory NHL including FL, MCL and MZL

DETAILED DESCRIPTION:
The study will conduct dose-finding. The dose-finding will be set as 3+3 design to seek candidates for optimal doses. Patients will receive study drugs to determine the MTD and/or OBD. In this study, OBD is defined as the most reasonable dose considering the benefit/risk ratio from available non-clinical and clinical data. The OBD will be determined based on available safety, PK/PD, and preliminary efficacy data, with a focus on identifying the dose that optimally balances clinical activity and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 to 80 years.
2. Patients must voluntarily agree to participate in the study and provide written informed consent prior to any study-related procedures.
3. Patients with histologically confirmed follicular lymphoma, mantle cell lymphoma or marginal zone lymphoma.
4. relapsed/refractory Patients who have received more than two prior lines of therapy.
5. Measurable disease based on Lugano classification.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
7. Adequate organ function including:

Exclusion Criteria:

1. Previous treatment with NB02 (poseltinib).
2. Patients who have experienced progression on BTKi mono or BTKi containing regimen (However, patients who discontinued treatment due to adverse-effect-related intolerance or for economic or social reasons remain eligible for enrollment).
3. Unable to take oral medication.
4. Inability to comply with study and follow-up procedures.
5. Concurrent use of other investigational drugs or enrollment in another clinical trial within 4 weeks prior to study drug administration.
6. Patients who have previously been treated with NB02 (poseltinib) or any other BTK inhibitors (e.g., ibrutinib, acalabrutinib, zanubrutinib).
7. Known HIV, HCV and HBV infection with active diseases

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD(maximum tolerated dose) or OBD(optimal biological dose) | Approximately 48 Months
  MTD(maximum tolerated dose) or OBD(optimal biological dose)
AEs | Approximately 48 Months
  AEs

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Ctrough | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) t1/2 | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) CL/F | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) Vz/F | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) Cmax | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) AUCtau | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Pharmacokinetic (PK) Tmax | Day 147
  Pharmacokinetic (PK) parameters from plasma samples
Overall response rate (ORR) | Approximately 48 Months
  To evaluate preliminary anti-tumor activity
Duration of response (DoR) | Approximately 48 Months
  To evaluate preliminary anti-tumor activity
Time to response (TTR) | Approximately 48 Months
  To evaluate preliminary anti-tumor activity
Progression-free survival (PFS) | Approximately 48 Months
  To evaluate preliminary anti-tumor activity
Overall Survival (OS) | Approximately 48 Months
  To evaluate preliminary anti-tumor activity

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seongnam
  - Catholic univ of Yeouido St Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan